CLINICAL TRIAL: NCT01804127
Title: Interim PET/CT Guided Cycle Numbers of R-CHOP in Patients With Diffuse Large B-cell Lymphoma: a Exploratory Phase II Study Study
Brief Title: Interim PET/CT Guided Cycle Numbers of R-CHOP in DLBCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ye Guo, Dr., Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LMTG 13-01
Record Dates: First submitted 2013-03-02; First posted 2013-03-05 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: DLBCL; R-CHOP; PET/CT
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — R-CHOP protocol; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- R-CHOP (Experimental): rituximab 375mg/m2 day 0, cyclophosphamide 750mg/m2 IV day 1, doxorubicin 50mg/m2 IV day 1, vincristine 1.4mg/m2 IV day1 (maximum: 2mg), prednisone 50mg PO days 1-5 twice per day
  Interventions: Drug: R-CHOP

INTERVENTIONS:
Drug: R-CHOP — rituximab 375mg/m2 day 0, cyclophosphamide 750mg/m2 IV day 1, doxorubicin 50mg/m2 IV day 1, vincristine 1.4mg/m2 IV day1 (maximum: 2mg), prednisone 50mg PO days 1-5 twice per day
  Other Names: mabthera

SUMMARY:
The aim of this study is to optimize the number of cycles of R-CHOP in patients with diffuse large B-cell lymphoma based on the interim results of PET/CT.

DETAILED DESCRIPTION:
R-CHOP is the standard regimen for patients with diffuse large B-cell lymphoma (DLBCL). However, the standard number of cycles is uncertain. Recently, interim PET/CT was found to predict prognosis in DLBCL. The hypothesis of this study is to optimize the number of cycles based on the interim results of PET/CT in order to avoid treatment exposure.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated diffuse large B-cell lymphoma
* Age range 18-80 years old
* Eastern Cooperative Oncology Group performance status 0-2
* Life expectancy of more than 3 months
* Adequate organ function

Exclusion Criteria:

* Primary or secondary central nervous system involvement
* Previous serious cardiac disease
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Pregnant or lactating women
* Serious uncontrolled diseases and intercurrent infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
3-year progression-free survival | 3 years

SECONDARY OUTCOMES:
Objective response rate | 6 months
3-year overall survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Jin J, Ji D, Xia Z, Xue K, Zhang Q, Liu Y, Cao J, Hong X, Gu JJ, Guo Y, Lv F. Four cycles of R-CHOP followed by two applications of rituximab based on negative interim PET/CT: an analysis of a prospective trial. BMC Cancer. 2022 Apr 13;22(1):403. doi: 10.1186/s12885-022-09486-4. PMID 35418080